CLINICAL TRIAL: NCT02440841
Title: Single Center, Open-Label, Single-Sequence, Within-Subject Study In Two Cohorts Of Healthy Male Subjects Comparing Single-Dose Pharmacokinetics Of Fedovapagon Alone And In Combination With A CYP3A4 Inhibitor, Itraconazole, Or A CYP3A4 Inducer, Rifampicin
Brief Title: Study in Healthy Male Subjects to Evaluate the Effect of Itraconazole and Rifampicin on the PK of Fedovapagon
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 483-010
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Nocturia
Keywords: VA106483; fedovapagon; drug-drug interaction; DDI; males; rifampicin; rifampin; itraconazole; CYP3A4; pharmacokinetics; PK
MeSH Terms: conditions — Nocturia | interventions — Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fedovapagon and itraconazole (Experimental): Two daily doses of fedovapagon and once daily doses of itraconazole
  Interventions: Drug: fedovapagon; Drug: Itraconazole
- fedovapagon and rifampicin (Experimental): Two daily doses of fedovapagon and once daily doses of rifampicin
  Interventions: Drug: fedovapagon; Drug: rifampicin

INTERVENTIONS:
Drug: fedovapagon
Drug: Itraconazole
  Arms: fedovapagon and itraconazole
Drug: rifampicin
  Arms: fedovapagon and rifampicin

SUMMARY:
The purpose of this study is to investigate the potential for co-administration of strong inhibitors or inducers of CYP3A4 to alter the pharmacokinetics of fedovapagon.

DETAILED DESCRIPTION:
Fedovapagon is a vasopressin V2 receptor agonist in development for the treatment of nocturia. Agonism of the V2 receptor, located in the collecting ducts of the kidney, leads to translocation of aquaporin channels and increased re absorption of water and anti-diuresis.

A number of drugs that are commonly co-prescribed in the population who may present for treatment of nocturia are inhibitors of CYP3A4, including diltiazem, verapamil, erythromycin and clarithromycin and may therefore impact the plasma levels of fedovapagon if co administered.

Conversely, concomitant intake of drugs that are potent CYP3A4 inducers may lead to lower than anticipated plasma concentrations of fedovapagon thus reducing the efficacy of fedovapagon. It is therefore important to assess the effect of CYP3A4 induction on the pharmacokinetic (PK) parameters of fedovapagon.

The study design uses itraconazole as a potent inhibitor of CYP3A4 and, in a separate cohort of subjects, rifampicin as a potent CYP3A4 inducer at doses intended to maximize the potential to demonstrate an interaction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males aged 18 to 45
* Have a body mass index between 18 and 29.9 kg/m2 (weight: ≥50 kg and ≤100 kg)
* No clinically significant medical history
* Ability to comply with the requirements of the study
* Provide written informed consent
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) should be below or equal to upper level of normal (ULN). Otherwise liver enzymes should show no clinical significant abnormalities. Total bilirubin should not exceed 1.5 x ULN. Liver enzymes will be re-tested only once before randomization if required.
* Be judged by the Investigator to be in good health based on medical history (in particular, no congestive heart failure, ischemic heart disease, valvular heart disease, significant pulmonary disease, renal failure, edematous disorder, liver disease, gastric disorders, porphyria, diabetes mellitus or hereditary disorders of carbohydrate metabolism), physical examination, vital sign measurements and laboratory safety tests
* Agree to refrain from the consumption of grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussels sprouts, mustard) and charbroiled meats containing products beginning 1 week prior to administration of the initial administration of trial drug, throughout the trial
* Use of any prescribed medication or St John's Wort within 14 days (or 5 half-lives if this is longer) or over-the-counter medication (except paracetamol) within 1 week of dosing. Specific medication not to be taken within 2 weeks of (before or after) administration of itraconazole is described in the Summary of Product Characteristic for Sempera®

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Plasma fedovapagon concentration in presence and absence of co-administered itraconazole or rifampicin | 10-12 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 10-12 days
Area under the plasma concentration curve versus time curve with extrapolation to infinity (AUC(0-infinity)) | 10-12 days
Number and type of adverse events | 12-14 days
Change from baseline in 12-lead ECG | 12-14 days
Change from baseline in vital signs and physical examination | 12-14 days
Change from baseline in laboratory assessments | 12-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Tshibuabua Kabasela, Study Director — Parexel
Locations (1):
- PAREXEL Early Phase Clinical Unit Berlin, Berlin, Germany